CLINICAL TRIAL: NCT04467814
Title: Out and About: Reablement for Older Adults in the Hospital Setting
Brief Title: Better Together: Reablement and Caregivers
Acronym: B2G
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-related issues had to change study design.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Maureen C. Ashe, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H20-01612
Record Dates: First submitted 2020-07-06; First posted 2020-07-13 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Older Adults; Sedentary Behavior; Physical Activity; Caregiver
Keywords: caregiver, patient, e-Course
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Better Together
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Better Together — Patient and caregiver dyads from both groups will receive usual care during hospitalization and following discharge. This will include a handout on strategies for safely remaining active.
  Caregiver participants in the intervention group will receive up to six telephone or video calls with the research assistant or Clinical Resource Therapist. Sessions will review the knowledge translation (KT) product with family members (~15 minutes), art goals, brainstorm strategies, and discuss setbacks. The calls with the caregiver may occur 1 to 2 times in the hospital, within one week of going home, and then in Months 2 and 3.
  Arms: Intervention
Behavioral: Usual Care — Patient and caregiver dyads from both groups will receive usual care during hospitalization and following discharge. This will include a handout on strategies for safely remaining active.
  Arms: Usual Care

SUMMARY:
Hospitalization creates opportunities for older adults to accumulate prolonged periods of sitting and lying (defined as sedentary behavior) which can result in mobility loss. We propose a Type 1 Hybrid Effectiveness-Implementation Trial with 1:1 randomization to test the effect of a caregiver intervention on older patients' physical activity at 3 months (home). We will recruit 61 patients and family caregivers from hospital units and follow them for 3 months; the primary outcome is patients' daily step count at 3 months.

ELIGIBILITY:
Inclusion Criteria: Older adults (60 years and older) with a recent hospitalization and their caregiver.

Exclusion Criteria: Caregivers and older adults with a dementia diagnosis, head injury, significant neurological impairment, or receive treatment for medical conditions that preclude exercising.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Veterans Rand-12 Quality of Life | baseline and 3 months
  12 item quality of life survey

SECONDARY OUTCOMES:
Daily minutes sedentary behavior | baseline to 3 months
  daily minutes of sedentary behavior measured with an activity monitor
Daily minutes of physical activity | baseline to 3 months
  daily minutes of physical activity measured with an activity monitor
Patient Assessment with Chronic Illness Care Survey | 3 months
  20-item survey with questions related to experience with hospitalization.
Brief Action Planning (BAP) | baseline and 3 months
  Goal setting
Action Plans behaviors | baseline and 3 months
  self-reported health behavior questions
Coping Plans | baseline and 3 months
  self-reported health behavior questions
Physical Activity Intentions | baseline and 3 months
  self-reported health behavior questions
Physical Activity Self-efficacy | baseline and 3 months
  self-reported health behavior questions
Physical Activity Risk Perceptions | baseline and 3 months
  self-reported health behavior questions
Physical Activity Outcome Expectancies | baseline and 3 months
  self-reported health behavior questions
Self-reported Habit Index | baseline and 3 months
  self-reported health behavior questions
Program implementation | baseline and 3 months
  Semi-structured interviews or focus groups with patients, caregivers, and heath providers to understand factors related program implementation.

OTHER OUTCOMES:
Steps per day | baseline to 3 months
  activity monitor
Falls | baseline to 3 months
  monthly falls diary
Falls Efficacy Scale International (FES-I) | baseline and 3 months
  16 questions related to falls self-efficacy. Scoring: minimum 16 (no falling concerns) to maximum 64 (high falling concern)
Brief Test of Adult Cognition by Telephone | baseline and 3 months
  cognitive test
Unified Theory of Acceptance and Use of Technology 2 Survey | baseline and 3 months
  self-report questions on perceptions of using technology

CONTACTS AND LOCATIONS:
Locations (1):
- The University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No